CLINICAL TRIAL: NCT02619006
Title: Effects of Placental Transfusion on Early Brain Development in Infants Born at Term: Follow-Up at 3 & 4 Years of Age
Brief Title: Infant Brain Study Follow-Up at 3 and 4 Years of Age
Status: Terminated | Type: Observational
Why Stopped: Lack of Funding
Sponsor: University of Rhode Island (Other)
Collaborators: Women and Infants Hospital of Rhode Island (Other); Brown University (Other)
Responsible Party: Principal Investigator, Judith S Mercer, Principal Investigator, University of Rhode Island
Other Study IDs: HU1112-086
Record Dates: First submitted 2015-11-23; First posted 2015-12-02 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-09

CONDITIONS: Iron Deficiency; Child Development
Keywords: Anemia, Iron-Deficiency; Myelination; Ferritin; Umbilical cord clamping; Umbilical Cord Milking; Placental Transfusion; Brain Development
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency; Fetofetal Transfusion | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immediate Cord Clamping: Healthy term infants who were previously randomized or assigned at birth to the control group known as immediate cord clamping. The cord was clamped and cut within10 seconds after birth.
- Delayed Cord Clamping or Cord Milking: Healthy term infants who were previously randomized or assigned at birth to the intervention group known as delayed cord clamping. The cord was clamped and cut at or beyond 300 seconds (5 mins). Cord milking (cord milked x 5) was used as a proxy for delayed cord clamping when there was a clinical situation of concern.
  Interventions: Other: Delayed Cord Clamping or Cord Milking

INTERVENTIONS:
Other: Delayed Cord Clamping or Cord Milking — Healthy term infants who were previously randomized or assigned at birth to the intervention group known as delayed cord clamping. The cord was clamped and cut at or beyond 300 seconds (5 mins). Cord milking (cord milked x 5) was used as a proxy for delayed cord clamping when there was a clinical situation of concern.
  Groups: Delayed Cord Clamping or Cord Milking

SUMMARY:
When immediate clamping of the umbilical cord (ICC) occurs at birth, 20 to 30% of the fetal-placental blood volume is left behind in the placenta. Preliminary results from our current study comparing effects of ICC versus placental transfusion from delayed cord clamping (DCC) show that infants who have DCC have higher ferritin levels at 4 months of age and more myelin in important regions of the brain. Our objective for this follow-up study is to see if the effects of placental transfusion persist to three and four years of age. The investigators plan to enroll only children who participated in the previous trial (Infant Brain Study/NCT01620008) at birth for assessments at three and four years of age. Assessments include MRIs and neurodevelopmental testing to examine cognitive, motor, visual, and behavioral outcomes.

The proposed research addresses two central questions regarding the potential benefits of DCC on brain myelin development in children who were born healthy at term: 1. Does DCC result in increased brain myelin deposition at three and four years of age? and 2) Are DCC, iron stores, and brain myelin content in infancy associated with improved cognitive, motor, and socio-behavioral outcomes at three and four years of age?

DETAILED DESCRIPTION:
The current obstetrical practice at birth in the United States is to cut and clamp umbilical cord of the infant immediately after birth. When immediate clamping occurs, 20 to 30% of the fetal-placental blood volume is left behind in the placenta. This blood contains enough iron-rich red blood cells to meet the infant's iron needs for the first 4 to 6 months of life. Delaying cord clamping has been shown to increase early iron stores without contributing to adverse outcomes. The investigators hypothesize that iron sufficiency is essential for long-term neurologic health. Iron deficiency in infancy adversely affects cognitive, motor, socio-emotional, and behavioral development. Human and animal studies have shown that inadequate iron stores in early infancy have an irreversible negative impact on the developing brain with deficits persisting even after iron levels have been restored by iron supplementation. Iron is an essential component of myelination which is critical for normal brain development and function. Myelination, which peaks during the first year of life, establishes and maintains efficient communication between the discrete regions of the brain.

The gap is that the effect of increased iron stores from delayed cord clamping on myelination and long-term neurodevelopment during childhood is unknown. Our hypothesis is that placental transfusion affects myelination and early childhood neurodevelopment in the following ways: 1) placental transfusion (delayed cord clamping or cord milking) leads to increased blood volume (BV) and red blood cell volume (RBCV) at birth; 2) increased RBCV results in more available iron for early body iron stores; 3) increased body iron stores provide essential iron supply for optimal brain myelination; 4) optimal myelination results in improved cognitive, behavioral and socio-emotional performance.

The main objective of this study is to conduct a prospective cohort study following the children enrolled in a previous randomized controlled trial (birth to 24 months) known as the Infant Brain Study. The purpose is to measure the effects of cord clamping time on the structure and function of the developing brain at three and four years of age. The investigators will use a non-invasive neuroimaging technique to measure myelin acquisition over time and conduct neurodevelopmental assessments and correlate the findings with early iron stores and long-term developmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Children who previously participated in the Infant Brain Study

Exclusion Criteria:

Ages: 30 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The eligible population includes 106 children who randomized in the controlled trial known as the "Effects of Placental Transfusion on Early Brain Development" (Infant Brain Study) (NCT01620008). The children were randomized to either immediate cord clamping or delayed cord clamping (or cord milking as a proxy for delayed clamping). The study population also includes a parallel preference group that self-selected cord clamping timing.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Brain myelination trajectory | 48 months of age
  Using MRI (McDespot technique) to map the myelin water volume fraction in brain

SECONDARY OUTCOMES:
Composite 48 Months of Age Neurodevelopmental Assessment | 48 months of age
  At 48 months of age using a composite of neurodevelopmental testing (i.e. Mullens Scales of Early Learning) and parent assessment questionaires (i.e. Child Behavior Checklist [CBCL]

CONTACTS AND LOCATIONS:
Overall Officials: Judith S Mercer, PhD, Principal Investigator — University of Rhode Island, Women and Infants Hospital of Rhode Island; Debra A Erickson-Owens, PhD, Principal Investigator — University of Rhode Island, Women and Infants Hospital of Rhode Island; Sean Deoni, PhD, Principal Investigator — Brown University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mercer JS, Erickson-Owens DA. Rethinking placental transfusion and cord clamping issues. J Perinat Neonatal Nurs. 2012 Jul-Sep;26(3):202-17; quiz 218-9. doi: 10.1097/JPN.0b013e31825d2d9a. PMID 22843002
- [Background] Erickson-Owens DA, Mercer JS, Oh W. Umbilical cord milking in term infants delivered by cesarean section: a randomized controlled trial. J Perinatol. 2012 Aug;32(8):580-4. doi: 10.1038/jp.2011.159. Epub 2011 Nov 17. PMID 22094494
- [Background] Deoni SC, Dean DC 3rd, Piryatinsky I, O'Muircheartaigh J, Waskiewicz N, Lehman K, Han M, Dirks H. Breastfeeding and early white matter development: A cross-sectional study. Neuroimage. 2013 Nov 15;82:77-86. doi: 10.1016/j.neuroimage.2013.05.090. Epub 2013 May 28. PMID 23721722
- [Result] Mercer JS, Erickson-Owens DA, Collins J, Barcelos MO, Parker AB, Padbury JF. Effects of delayed cord clamping on residual placental blood volume, hemoglobin and bilirubin levels in term infants: a randomized controlled trial. J Perinatol. 2017 Mar;37(3):260-264. doi: 10.1038/jp.2016.222. Epub 2016 Dec 8. PMID 27929530
- [Result] Mercer JS, Erickson-Owens DA, Deoni SCL, Dean DC 3rd, Collins J, Parker AB, Wang M, Joelson S, Mercer EN, Padbury JF. Effects of Delayed Cord Clamping on 4-Month Ferritin Levels, Brain Myelin Content, and Neurodevelopment: A Randomized Controlled Trial. J Pediatr. 2018 Dec;203:266-272.e2. doi: 10.1016/j.jpeds.2018.06.006. Epub 2018 Jul 6. PMID 30473033